CLINICAL TRIAL: NCT00622141
Title: Bioequivalence Study of Generic GPO Saquinavir and Norvir® Versus Invirase® and Norvir® in Thai Healthy Volunteers
Brief Title: Bioequivalence Study of Generic GPO Saquinavir and Norvir® Versus Invirase® and Norvir®
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was never started because the sponsor decided not to manufacture the investigational product.
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government)
Responsible Party: Professor Kiat Ruxrungtham, HIV-NAT
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HIV-NAT 038
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: bioequivalence; ritonavir boosted generic GPO saquinavir; saftey; pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Day 1: receive a single dose of Invirase®/Norvir® 1,000 mg / 100mg 7-day washout period will follow. Day 8: take generic GPO squinavir/Norvir
  Interventions: Drug: generic GPO saquinavir and novir vs invirase and norvir
- B (Active Comparator): Day 1: take generic GPO squinavir/Norvir 7-day washout period will follow. Day 8: receive a single dose of Invirase®/Norvir® 1,000 mg / 100mg
  Interventions: Drug: generic GPO saquinavir and novir vs invirase and norvir

INTERVENTIONS:
Drug: generic GPO saquinavir and novir vs invirase and norvir — Norvir® 100mg capsules, Invirase® 1,000 mg capsules Generic GPO Saquinavir 1,000 mg capsules For phase 1 and 2 - At day 1 subjects of group A will receive a single dose of Invirase®/Norvir® 1,000 mg / 100mg, while group B will receive generic GPO saquinavir / Norvir® 1,000 mg / 100mg as single dose. The same day the first 24 hr PK curve will be done. After this, a 7-day washout period will follow. At day 8 group A will take generic GPO saquinavir / Norvir® and Group B will take Invirase®/Norvir®. At this day, the second 24 hr PK curve will be done

SUMMARY:
The previous two studies of generic GPO saquinavir failed to prove bioequivalence. In this study the bio-equivalence will be investigated in healthy Thai volunteers, to see whether the generic GPO saquinavir shows bioequivalence when boosted with Norvir®. If the generic formulation is bioequivalent subsequent studies may follow in HIV-1 positive patients.

DETAILED DESCRIPTION:
The primary objective is to establish bioequivalence of "ritonavir boosted generic GPO saquinavir", with Invirase® and Norvir® as the reference drug.

The secondary objective is to evaluate the short-term tolerability and safety profiles of generic saquinavir in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy male 18-45 years old
* Documented negative test for HIV-1 infection < 1 wk prior to start of study and with no risk of HIV exposure in the last 6 months
* BMI 18-25
* Normal physical examination
* Normal CBC, BUN, Cr, AST, ALT, Total bilirubin, no evidence of active or chronic HBV or HCV infection

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to the drug or chemically related compounds or excipients, which may be employed in the study.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the study and the procedures required.
* Participation in a drug study within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose.
* Use of concomitant medication
* Smoke cigarettes not more than 10 cigarettes a day.
* Drink alcohol not more than 2 units a day.
* Discontinue smoking and alcohol for at least 1 month before enrollment.
* Take other medication regularly
* Involvement in any drug addiction.
* Heart disease, hypertension, liver disease, kidney disease, GI disease, allergic disease or other diseases which may interfere with the PK of study drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To establish bioequivalence of ritonavir boosted generic GPO saquinavir generic, with Invirase® and Norvir® as reference drug. | 8 days

SECONDARY OUTCOMES:
The secondary objective is to evaluate the short-term tolerability and safety profiles of generic saquinavir in healthy male volunteers. | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org